CLINICAL TRIAL: NCT00999960
Title: A Prospective Randomized Study to Evaluate the Clinical Impact of a Laparoscopic Radical Prostatectomy Online Simulator
Brief Title: Study to Evaluate the Clinical Impact of a Laparoscopic Radical Prostatectomy Simulator
Acronym: PERLE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of sponsor
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOR 07074-NI07008
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Prostatic Neoplasms; Cancer of Prostate; Prostate Cancer; Prostate Neoplasms
Keywords: Laparoscopy; Prostate; Cancer; Learning; Simulation; Simulator
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: without simulator (Active Comparator): without simulator
  Interventions: Procedure: Laparoscopic Radical Prostatectomy (without a simulator)
- 2: with simulator (Experimental): with simulator
  Interventions: Procedure: Laparoscopic Radical Prostatectomy (with a simulator)

INTERVENTIONS:
Procedure: Laparoscopic Radical Prostatectomy (without a simulator) — without simulator
  Arms: 1: without simulator
Procedure: Laparoscopic Radical Prostatectomy (with a simulator) — Learning with a simulator
  Arms: 2: with simulator

SUMMARY:
To evaluate the clinical impact of an online video simulator during the learning period of laparoscopic radical prostatectomy.

DETAILED DESCRIPTION:
Objectives: To compare two different approaches in learning laparoscopic radical prostatectomy , with or without using an online video simulator Design : Prospective randomized multicentric study

Methods: 20 surgeons considered as naive concerning their experience in laparoscopic radical prostatectomy will be randomized into two groups :1 group will use the online video simulator, 1 group will use usual learning methods except the online video simulator.

All procedures will be recorded from the beginning till the end.A video review will be preformed concerning all the videos in order to identify the total operative time and time to perform each one of the operative steps of the procedure.Clinical , biological and histological data will be collected in order to compare the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon beginning his clinical experience in laparoscopic radical prostatectomy and having performed less then 30 procedures before being enrolled in the study
* Surgeon who intends to begin laparoscopic radical prostatectomy clinical practice
* Surgeons who usually perform enough cases to enroll at least 10 patients during the study inclusion time

Exclusion Criteria:

* Surgeon who does not have access to high speed internet (>1024 Ko/s)
* Surgeons who do not intend to begin laparoscopic radical prostatectomy in his clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Operative time to perform the complete procedure | during the procedure

SECONDARY OUTCOMES:
Operative time to complete each step of the procedure | each step of the procedure
Intraoperative bleeding | during the procedure
Transfusion rate | Hospital stay
Complication rate | during the procedure
Conversion rate | during the procedure
Quantity of liquid obtained in drains | during the hospitalization
Duration of urethral stenting | during the hospitalization
Reintervention rate | during the patient participation
Duration of hospital stay | during the patient participation
Positive surgical margin | during the procedure
PSA value | at 3,6 and 12 months after the procedure
Continence rate | at 3, 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: DESGRANDCHAMPS François, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HOPITAL SAINT-LOUIS Service d'urologie, Paris, France